CLINICAL TRIAL: NCT00910585
Title: Phase 4 Study of Case Management and Environmental Control in Asthma
Brief Title: Coaching in Childhood Asthma
Acronym: Coach
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Robert C. Strunk, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ES08711
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Asthma
Keywords: childhood; asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active coaching (Experimental): Telephone and in person coaching
  Interventions: Behavioral: Coaching, providing social support
- Usual care (Active Comparator): Return to PCP for usual care
  Interventions: Behavioral: Coaching, providing social support

INTERVENTIONS:
Behavioral: Coaching, providing social support — Active telephone and in person coaching

SUMMARY:
Asthma among low-income, minority children remains a prime example of health disparities that are resistant to change. Demonstrations of reductions in disproportionate hospitalizations in controlled trials are limited. We performed a controlled clinical trial of an Asthma Coach to reduce hospitalizations among low-income, African American children.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of children with asthma 2-8 years of age and hospitalized for an acute exacerbation, with Medicaid insurance, and living in St. Louis City

Exclusion Criteria:

* Other respiratory disease present

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 1997-01; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Rehospitalization | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Strunk, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States